CLINICAL TRIAL: NCT06278792
Title: Readily Available Urinary Sodium Analysis in Patients With Acute Decompensated Heart Failure
Acronym: EASY-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z-2021104
Record Dates: First submitted 2024-02-08; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Acute Decompensated Heart Failure
Keywords: acute decompensated heart failure; natriuresis; nurse-led; diuretic therapy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The EASY-HF study was a single-centre, randomized, open-label study comparing standard of care (SOC) diuretic management at the treating physician's discretion with a nurse-led natriuresis-guided protocol in patients with ADHF.
Who Masked: Participant, Care Provider
Masking Description: All physicians were blinded for the spot urinary sodium measurements. Additionally, while urine was collected for the first 48 h in both groups, the analysis was only performed afterwards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): 48 hour diuretic management at the treating physician's discretion
  Interventions: Procedure: Standard of Care
- Intervention (Experimental): 48-hour nurse-led natriuresis-guided protocol
  Interventions: Procedure: Diuretic protocol

INTERVENTIONS:
Procedure: Diuretic protocol — Nurse-led natriuresis-guided protocol based on a bedside urinary sodium result
  Arms: Intervention
Procedure: Standard of Care — Diuretic therapy at the discretion of the physician
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to compare physician-guided (SOC) versus nurse-led natriuresis-guided diuretic therapy in patients with acute decompensated heart failure (ADHF). The main questions it aims to answer are:

* difference in natriuresis and diuresis
* feasibility of the protocol.

Participants will be asked to gather two 24 h urine collections.

Researchers will compare SOC versus nurse-led diuretic titration to see if there is a difference in natriuresis after 48 hours.

DETAILED DESCRIPTION:
The EASY-HF study was a single-centre, randomized, open-label study comparing standard of care (SOC) diuretic management at the treating physician's discretion with a nurse-led natriuresis-guided protocol in patients with ADHF. A bedside sensor was used to measure the urinary sodium content.The primary endpoint was total natriuresis after 48 hours. Secondary endpoints included safety profile and user-friendliness of both the protocol and the point-of-care sensor.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Provide written informed consent
* Hospital admission with signs and symptoms of congestion warranting intravenous decongestive therapy
* Congestion score of at least 2 based upon the presence of edema, pleural effusion, or ascites
* N-terminal pro-B-type natriuretic peptide (NT-proBNP) level of at least 500 ng per litre (800 ng per litre in case of atrial fibrillation)

Exclusion Criteria:

* Patients unable to collect a 48h-urine collection
* Estimated GFR below 20 ml/min/1.73m^2
* Concomitant diagnosis of an acute coronary syndrome
* Need for inotropic or vasopressor support
* Ventricular assist device
* Renal replacement therapy
* Treatment with intravenous loop diuretics > 80mg furosemide or an equivalence of another loop diuretic (40mg furosemide = 1mg bumetanide) during the index hospitalization and prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Urinary sodium excretion after 48 hours | 48 hours
  Total natriuresis after 48 hours (mmol)

SECONDARY OUTCOMES:
Urinary output after 48 hours | 48 hours
  Total diuresis after 48 hours (ml)
Urinary sodium excretion on daily base | 24 hours
  Total natriuresis (mmol) during the first and second 24 h
Urinary output on daily base | 24 hours
  Total diuresis during the first and second 24 h
Achievement of decongestion | 48 hours
  Congestion score of no more than trace edema (score < 2) after 48 hours of diuretic treatment. Minimum score 0 (decongested), maximum score 10 (severe congested)

OTHER OUTCOMES:
Diuretic dose | 48 hours
  Dose of loop diuretics and other diuretic agents administered
User-friendliness device and protocol | 180 days
  Questionnaire for the nursing staff with regard to user-friendliness of device and diuretic protocol (1 (totally disagree) to 10 (completely agree))
Weight | 48 hours
  Body weight change
Number of participants with need for heart failure rehospitalization | 180 days
  Heart failure rehospitalization during the first 180 after start of the study
Rate of all-cause mortality | 180 days
  All-cause mortality during the first 180 after start of the study
Length of hospital stay | 180 days
  The time frame between hospital admission and discharge will be calculated
Number of participants with severe hypotension | 48 hours
  systolic blood pressure below 85mmHg
Number of participants with abnormal blood parameters | 3-day follow-up
  Any abnormal laboratory parameters in the blood (electrolytes, renal function) during a 3 day follow-up will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Mullens, MD PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg AV, Genk, Limburg, Belgium